### INFORMED CONSENT FORM

**Study Title:** The Effect of a Micro-Appreciation Intervention (Three-Things Journal Application) on Caregiver Burden, Family Functioning, and Happiness Levels for Mothers of

Children With Autism Spectrum Disorder: An Experimental Study

NCT Number: NCTXXXXXXX Document Date: August 1, 2025

#### **Informed Consent Statement**

This study has received written approval from the Institutional Review Board of Batman University Non-Interventional Clinical Research Ethics Committee. We invite you to voluntarily participate in this research.

Participation is completely optional, and you have the right to withdraw at any time without any consequences.

## **Purpose of the Study**

This study aims to investigate the effects of a micro-appreciation intervention (Three-Things Journal Application) on caregiver burden, family functioning, and happiness levels.

## **What Participation Involves**

If you agree to participate:

- You will be asked to use the Three-Things Journal Application for a specific period.
- You will complete questionnaires measuring caregiver burden, family functioning, and happiness levels.

## **Risks and Benefits**

During the study, you may experience emotional reactions while reflecting on your caregiving experience. If you feel any discomfort, you may stop at any time.

### **Confidentiality**

All information will be kept confidential and will only be used for research purposes.

# **Voluntary Participation**

You may refuse to participate or withdraw at any time without providing a reason or facing any negative consequences.

If you agree to participate, please sign below. You will receive a copy of this form.

| Participant Information and Consent | |
|-------------------------------------|---------------|
| Participant's Full Name: | |
| Address: | |
| Phone Number: | |
| Signature: | Date://2025 |
| Researcher Information | |
| Researcher's Full Name and Title: | |
| Institution / Address: | |
| Phone Number: | |
| Signature: | Date: / /2025 |